CLINICAL TRIAL: NCT06548217
Title: An Open-label, Uncontrolled, Phase I Study of ONO-4538HSC in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of ONO-4538HSC in Subjects With Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538HSC-01; jRCT2011230059 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ONO-4538HSC (Experimental)
  Interventions: Drug: ONO-4538HSC

INTERVENTIONS:
Drug: ONO-4538HSC — ONO-4538HSC will be administered subcutaneously once every 4 weeks.

SUMMARY:
This is a multicenter, open-label, uncontrolled, phase I study to evaluate the tolerability, safety, pharmacokinetics, and efficacy of ONO-4538HSC administered subcutaneously in participants with advanced or metastatic solid tumors. This study consists of the tolerability confirmation part to determine the recommended dose for Japanese participants by evaluating the DLTs and the expansion part to evaluate the safety and pharmacokinetics and to explore the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with advanced or metastatic solid tumors
2. Patients have an ECOG performance status of 0 to 1
3. Patients with a life expectancy of at least 3 months

   [Tolerability confirmation part]
4. Patients who are refractory or intolerant to standard therapy or for whom no standard therapy is available

   [Expansion part]
5. Patients who are refractory or intolerant to standard therapy, or for whom no standard therapy is available, or for whom monotherapy with intravenous nivolumab is indicated according to the package insert

Exclusion Criteria:

1. Patients with a complication or history of severe hypersensitivity to any antibody product
2. Patients with severe complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 28 days
Adverse event (AE) | UP to 100 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics（serum concentration of Nivolumab） | Up to Cycle25 (each cycle is 28 days) and Post-treatment observation phase (28 days after the end of treatment phase)

OTHER OUTCOMES:
Overall response rate (ORR) | Through study completion, an average of 6 months
Disease control rate (DCR) | Through study completion, an average of 6 months
Overall survival (OS) | Through study completion, an average of 6 months
Progression-free survival (PFS) | Through study completion, an average of 6 months
Duration of response (DOR) | Through study completion, an average of 6 months
Time to response (TTR) | Through study completion, an average of 6 months
Best overall response (BOR) | Through study completion, an average of 6 months
Percentage of change in the sum of tumor diameters of target lesions | Through study completion, an average of 6 months
Maximum percent change in the sum diameters of the target lesions | Through study completion, an average of 6 months
Anti-Nivolumab antibody | Up to Cycle25 (each cycle is 28 days) and Post-treatment observation phase (28 days after the end of treatment phase)
Anti-rHuPH20 antibody | Up to Cycle25 (each cycle is 28 days) and Post-treatment observation phase (28 days after the end of treatment phase)

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (8):
- Japan (8):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No